CLINICAL TRIAL: NCT04932343
Title: Comparison of Genomic and Transcriptomic Patterns Between the Circulating Tumor Cells and Metastatic Tumor Cells, and Their Specific Relevance to Circulating Tumor DNAs: Quest for Any Distinct or Complementary Roles of CTCs and ctDNAs to Understand the Metastasis in Advanced NSCLC
Brief Title: Comparison of Genomic and Transcriptomic Patterns Between CTC and Metastatic Tumormetastatic Tumor
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: CytoGen, Inc. (Industry); UNIST (Ulsan National Institute of Science and Technology) (Unknown)
Responsible Party: Principal Investigator, Jhingook Kim, MD, Professor, Samsung Medical Center
Other Study IDs: IRB 2019-07-101
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: NSCLC Stage IV; NSCLC Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cohort study — no intervention

SUMMARY:
This study aims to understand the metastasis in advanced NSCLC through comparing genomic and transcriptomic patterns between the circulating tumor cells and metastatic tumor cells by single cell sequencing analysis.

ELIGIBILITY:
Inclusion Criteria:

* All subjects need to sign the informed consent form
* All subjects have non-small cell lung cancer which suspected on chest CT or confirmed pathologically preoperatively
* Treatment naïve advanced lung cancer (including extensive stage IIIb and stage IV)
* Patients who were suitable to provide enough metastatic tumor tissue and blood (30ml) for the single cells sequencing

Exclusion Criteria:

* Patients with previous history of lung cancer
* Have been undergone chemotherapy or radiotherapy due to non-small call lung cancer
* Have been diagnosed any type of cancer other than cancer of skin, thyroid, uterine cervix within 5 years before enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment naïve stage III-IV non-small cell lung cancer who undergoing surgery for any intent
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The gene expression and the cell population | 3 year
  Methods for the single cell RNA sequencing and whole exome sequencing of the tumor cells With the tissue biopsied specimens, scRNAseq (by 10X Genomics platform) and whole exome seq will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Jhingook Kim, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided